CLINICAL TRIAL: NCT04265261
Title: A Randomized, Double-Masked, 48-Week, Parallel-Group, Placebo-Controlled, Proof-of-Concept Study to Investigate the Efficacy and Safety of RG7774 in Patients With Diabetes Mellitus Type 1 or Type 2 With Treatment-Naive Diabetic Retinopathy
Brief Title: A Study to Investigate the Efficacy and Safety of RG7774 in Patients With Diabetes Mellitus Type 1 or Type 2 With Treatment-Naive Diabetic Retinopathy
Acronym: CANBERRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP41321; 2019-002067-10 (EudraCT Number)
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Placebo Comparator): Participants will receive an oral dose of placebo matched to RG7774 once daily (QD)
  Interventions: Drug: Placebo
- Group B (Experimental): Participants will receive a low oral dose of RG7774 QD
  Interventions: Drug: RG7774
- Group C (Experimental): Participants will receive a high oral dose of RG7774 QD
  Interventions: Drug: RG7774

INTERVENTIONS:
Drug: Placebo — Participants will receive oral placebo matched to RG7774
  Arms: Group A
Drug: RG7774 — Participants will receive oral RG7774
  Arms: Group B; Group C

SUMMARY:
The study's main purpose is to asses the safety, tolerability, and effect of oral administration of RG7774 on the severity of diabetic retinopathy (DR) in participants with moderately severe to severe non-proliferative diabetic retinopathy (NPDR) and good vision.

ELIGIBILITY:
Inclusion Criteria

* Able and willing to provide written informed consent and to comply with the study protocol according to International Conference of Harmonization (ICH) and local regulations
* Male and female patients of at least 18 years of age
* Treatment naïve with moderately severe to severe NPDR defined as ETDRS DRSS 47 or 53
* Patients are eligible with and without DME in either eye
* BCVA score at screening of at least 70 letters in study eyes without DME and at least 75 letters in case DME is present
* Clear ocular media and adequate pupillary dilation to allow acquisition of good quality retinal images.
* Diagnosis of diabetes mellitus (DM) type 1 or type 2
* Hemoglobin A1c (HbA1c) </= 12%.
* A female is eligible to participate if she is not pregnant, not breastfeeding

Exclusion Criteria

Ocular criteria for study eye:

* Prior treatment for DR or other retinal diseases with any approved or investigational therapy, including but not limited to intravitreal steroids, intravitreal anti-VEGF, light therapy, periocular pharmacological intervention, and laser (e.g. focal, grid, micropulse, or pan-retinal)
* Uncontrolled glaucoma
* Any concurrent intraocular condition (e.g. retinal detachment, dense cataract, epiretinal membrane with traction, or vitreomacular traction, etc.) that in the opinion of the Investigator could reduce the potential for improvement, require medical surgical intervention or may confound the visual and functional assessment and interpretation of study results

Concurrent ocular conditions in either eye:

* Any active ocular infection
* Any active intraocular inflammation

General Criteria:

* Previous systemic use of anti-VEGF drugs within 6 months prior to screening
* Complications of diabetes such as end-stage renal disease or liver disease
* Currently untreated diabetes mellitus or previously untreated patients who initiated oral or injectable anti-diabetic medication within 3 months prior to screening
* Uncontrolled blood pressure ([BP] defined as systolic > 180mmHg and/or diastolic >100 mmHg while patient at rest)
* History of concurrent cardio-vascular disease not considered well controlled by the Investigator
* Any major illness or major surgical procedure within one month before screening
* History of or currently active other diseases, metabolic dysfunction, physical examination finding, malignancies not considered cured, or clinical laboratory findings giving reasonable suspicion of a condition that contraindicated the use of the investigational medicinal drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications in the opinion of the investigator
* Known hypersensitivity to any of the excipients of the drug used, fluorescein dye or dilating eye drops
* Use of systemic medications known to be toxic to the lens, retina or optic nerve (e.g., deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazines and ethambutol) used during the 6-month period prior to screening or likely need to be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (68):
- United States (37):
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retina Associates Tucson, Tucson, Arizona
  - Win Retina, Arcadia, California
  - Global Research Management, Glendale, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Retina Consultants of Southern Colorado PC, Colorado Springs, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Rand Eye, Deerfield Beach, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Medeye Associates, Miami, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Retina Associated Ltd, Elmhurst, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Deep Blue Retina PLLC, Southaven, Mississippi
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Velocity Clinical Research, East Syracuse, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Charlotte Eye Ear Nose and Throat Associates, Charlotte, North Carolina
  - EyeHealth Northwest, Portland, Oregon
  - Erie Retinal Surgery, Erie, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Retinal Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
- Australia (4):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
- Poland (5):
  - Centrum Medyczne Julianow; Zeglarska, ?ód?
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - Centrum Medyczne UNO-MED, Krakow
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
  - LensClinic, Rybnik
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Klinika Oftalmológie LFUK a UNB, Bratislava
  - O?ná klinika UNB a SZU, Bratislava
  - 3F s.r.o, Košice
  - Fakultna nemocnica Trencin, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina; Ocne oddelenie, Žilina
- Spain (8):
  - Hospital Universitari de Bellvitge; Servicio de Oftalmologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Dos de Maig, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Clinica Barraquer, Barcelona
  - Pio del Rio Hortega University Hospital, Valladolid
  - Miguel Servet University Hospital, Zaragoza
- United Kingdom (7):
  - Royal Victoria Hospital; Outpatients Department, Belfast
  - Colchester General Hospital, Colchester, Essex
  - Royal Surrey County Hospital; Eye Clinic Research office, Guildford
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Royal Liverpool University Hospital, Liverpool
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Armendariz BG, Luhman UFO, Berger B, Hernandez-Sanchez J, Bogman K, Mitrousis N, Wollenhaupt M, Kent D, Wenzel A, Fauser S. CANBERRA: A Phase II Randomized Clinical Trial to Test the Therapeutic Potential of Oral Vicasinabin in Diabetic Retinopathy. Ophthalmol Sci. 2024 Nov 8;5(2):100650. doi: 10.1016/j.xops.2024.100650. eCollection 2025 Mar-Apr. PMID 39802207

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received an oral dose of placebo matched to RG7774 once daily (QD)
- Vicasinabin 30 mg QD: Participants received 30 mg of oral RG7774 QD
- Vicasinabin 200 mg QD: Participants received 200 mg of oral RG7774 QD
Period: Overall Study
Arm/Group | Placebo | Vicasinabin 30 mg QD | Vicasinabin 200 mg QD
Started | 47 | 48 | 44
Completed | 37 | 43 | 36
Not Completed | 10 | 5 | 8
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 3
Not completed — Non-Compliance with Study Drug | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vicasinabin 30 mg QD | Vicasinabin 200 mg QD | Total
Number analyzed (Participants) | 47 | 48 | 44 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (9.3) | 57.3 (10.0) | 56.5 (10.5) | 57.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 16 | 51
  Male | 30 | 30 | 28 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 18 | 15 | 47
  Not Hispanic or Latino | 32 | 30 | 29 | 91
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 0 | 4 | 9
  White | 40 | 46 | 35 | 121
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With >/= 2-Step Improvement in the Early Treatment Diabetic Retinopathy Study (ETDRS) DR Severity Scale (DRSS) From Baseline at Week 36 Measured in the Study Eye
Description: The ETDRS DRSS is a standardized grading test to measure diabetic retinopathy progression, where higher scores indicate a higher risk of vision loss. The DRSS ranges from level 10 (no diabetic retinopathy) to level 85 (advanced diabetic retinopathy)
Time Frame: Week 36
Population: The mITT population is defined as all participants who give informed consent, are randomized, and receive at least one dose of study treatment (active or placebo). For the mITT population, data were analyzed according to the treatment participants were randomized to.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Vicasinabin 30 mg QD | Vicasinabin 200 mg QD
Number analyzed (Participants) | 38 | 42 | 35
Percentage of participants | 7.89 [2.72 to 20.8] | 9.52 [3.77 to 22.07] | 5.71 [1.58 to 18.61]
Statistical Analysis 1: Comparison: Placebo vs Vicasinabin 30 mg QD; Test type: Superiority; p = 0.8586, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.19, 95% CI 2-sided [-11.86 to 14.23]
Statistical Analysis 2: Comparison: Placebo vs Vicasinabin 200 mg QD; Test type: Superiority; p = 0.6388, Cochran-Mantel-Haenszel; Risk Difference (RD) = -2.93, 95% CI 2-sided [-15.18 to 9.31]

2. Secondary Outcome: Time-to-Event for Vision-Threatening DR in the Study Eye
Description: Vision-threatening DR was defined as anterior segment neovascularization (ASNV), new proliferative diabetic retinopathy (PDR), new diabetic macular edema (DME), and pre-existing DME requiring treatment. Time-to-event was defined as the time where 50% of the population develops a DR vision-threatening event.
Time Frame: Up to Day 277
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Vicasinabin 30 mg QD | Vicasinabin 200 mg QD
Number analyzed (Participants) | 47 | 48 | 43
Days | NA [257.0 to NA] — NA indicates that either the Kaplan-Meier percentile time has not been achieved or that the percentile is at a boundary of the observed range and no upper or lower 95% CI can be found due to insufficient sample size. | 267.0 [254.0 to NA] — NA indicates that either the Kaplan-Meier percentile time has not been achieved or that the percentile is at a boundary of the observed range and no upper or lower 95% CI can be found due to insufficient sample size.. | NA [260.0 to NA] — NA indicates that either the Kaplan-Meier percentile time has not been achieved or that the percentile is at a boundary of the observed range and no upper or lower 95% CI can be found due to insufficient sample size..

3. Secondary Outcome: Incidence of New Anterior Segment Neovascularization (ASNV), New Proliferative Diabetic Retinopathy (PDR), New Diabetic Macular Edema (DME), and Pre-Existing DME Requiring Intervention in the Study Eye
Description: This is a descriptive summary of the incidence of new ASNV, new PDR, new DME, and pre-existing DME, all of which indicate disease progression. Each row presents the proportion of participants amongst the overall population for each event.
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Vicasinabin 30 mg QD | Vicasinabin 200 mg QD
Number analyzed (Participants) | 47 | 48 | 43
Percentage of participants
  New ASNV | 0 [0.0 to 9.4] | 0 [0.0 to 9.2] | 0 [0.0 to 10.2]
  New PDR | 0 [0.0 to 9.4] | 6.3 [1.6 to 18.2] | 0 [0.0 to 10.2]
  New DME | 0 [0.0 to 9.4] | 4.2 [0.7 to 15.4] | 0 [0.0 to 10.2]
  Pre-existing DME requiring treatment | 4.3 [0.7 to 15.7] | 10.4 [3.9 to 23.4] | 6.8 [1.8 to 20.1]

4. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye at Week 36
Description: BCVA was measured by a qualified VA examiner prior to pupil dilation using modified ETDRS Charts 1, 2, and R. The adjusted mean is reported for each group.
Time Frame: Baseline; Week 36
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of letters
Arm/Group | Placebo | Vicasinabin 30 mg QD | Vicasinabin 200 mg QD
Number analyzed (Participants) | 47 | 48 | 43
Number of letters | 0.12 (0.747) | -0.45 (0.697) | -0.22 (0.744)

5. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Up to 1 year (baseline through follow-up period)
Population: The Safety population is defined as all participants who give informed consent, receive at least one dose of study medication (active or placebo) and were grouped according to the actual treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Vicasinabin 30 mg QD | Vicasinabin 200 mg QD
Number analyzed (Participants) | 47 | 48 | 43
Percentage of participants | 72.3 | 64.6 | 81.4

ADVERSE EVENTS:
Time Frame: Up to 1 year (baseline through follow-up period)
Description: All-cause mortality includes the entire study population. SAE and NSAE reporting includes the safety population, which included all participants who gave informed consent and received at least one dose of study medication. Participants in the safety population were grouped according to the actual treatment received.
Arm/Group | Placebo | Vicasinabin 30 mg QD | Vicasinabin 200 mg QD
All-Cause Mortality (participants affected / at risk) | 1/47 | 0/48 | 0/44
Serious Adverse Events (participants affected / at risk) | 8/47 | 3/48 | 5/43
Other Adverse Events (participants affected / at risk) | 13/47 | 21/48 | 15/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Vicasinabin 30 mg QD (N=48) | Vicasinabin 200 mg QD (N=43)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Vicasinabin 30 mg QD (N=48) | Vicasinabin 200 mg QD (N=43)
Diabetic retinal oedema (Eye disorders) | 3 (3) | 8 (13) | 6 (7)
Diabetic retinopathy (Eye disorders) | 3 (3) | 5 (5) | 1 (2)
Vitreous haemorrhage (Eye disorders) | 1 (2) | 3 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (4) | 3 (3) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT04265261/Prot_SAP_000.pdf